CLINICAL TRIAL: NCT03234868
Title: Benefit of the Digital Workflow for Screw-retained Single Implant Restorations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Dr. France LAMBERT, Prof., University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H2015-4
Record Dates: First submitted 2017-04-13; First posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Optical impression (Experimental): The optical impression system used for the study is TRIOS (3 shape). First of all, the operators in charge of taking the digital impressions are going to get trained prior the study and will calibrate (learning curve). MIS Scan bodies will be placed on the multi-unit plaforms, an x-ray will be taken in order to check the fit) and the impression will be realised following the instruction given by the system (first the maxillary and mandibular impressions followed by the bite registration). Shade will be chosen using VITA toothguide 3D master (to pick the right zirconia shade).
  Interventions: Device: Impression procedure
- Conventional impression (Active Comparator): Once the impression coping is placed on the multi-unit plaform, the fit will be checked with an intra-oral X-ray. The impressions will be made with medium viscosity silicon. As a second step, alginate antagonist impression will be done. Bite will not be recorded (single tooth missing). The two impressions will be placed in a hermetic plastic bag and send to lab. Shade will be chosen using VITA toothguide 3D master.
  Interventions: Device: Impression procedure
- Digital workflow (Experimental): The implant crowns issued from digital impressions will be done according a cast less / full digital workflow. The STL files collected from the TRIOS will be sent directly to the lab. The designing of the full zirconia crowns will be performed in the TRIOS 3SHAPE program. The resulting files will be sent to the CAM unit production (Amman Girrbach milling machine & MAZAK CNC machine: Mcenter to be specify (Berlin or Israel) to be milled (milled & sintered only) considering the direct adaption for a Multi-Unit connection. A superficial make-up will be done on the monolithic crown in the lab. And finally, the products will be delivered to the dentist.
  Interventions: Device: Crown manufacturing procedures
- Conventional workflow (Active Comparator): The implant crowns issued from conventional impressions will be realised by sending the impressions to the lab (Mirko Picone). The lab will pour the impressions in dental stone (class 4 scannable without powdering: extra hard and scanning powder included). Then, the technician will realize a mock-up of the crown's framework on a temporary abutment in DuraLay Resin.
  The mock up will be scanned with ZIRKONZAHN scanner (or equivalent) and send this information to a central fabrication facility for milling (Amman Girrbach milling machine & MAZAK CNC machine:
  Mcenter: to be specify (Berlin or Israel). The lab technician will get the Zi framework back and will apply veneer ceramic.
  Interventions: Device: Crown manufacturing procedures

INTERVENTIONS:
Device: Impression procedure — Each patient will go through both type of impression during single appointment: first the digital impression and then the conventional one (to avoid residual impression materials for the optical impressions). The time necessary for each procedure will be recorded.
  Arms: Conventional impression; Optical impression
Device: Crown manufacturing procedures — Test and control implant crowns will be screw-retained on a multi-unit abutment. The conventional crown will be made of a Zirconia framework veneered with cosmetic ceramics directly screwed on the multi-unit platform (no titanium base). The experimental crown will be made in full zirconia and designed in the TRIOS software.
  Arms: Conventional workflow; Digital workflow

SUMMARY:
The aim of this research project is emphasize the benefit of the digital workflow compared to conventional impressions and crown processing with standard la procedures. The objectives of the present study are to measure and compare the global cost, the time spent in the dental chair and in the lab and the fit of both digital and conventional workflow. Additionally, patient centered outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have voluntarily signed the informed consent form before any study related action
* Age: 18 with one or more missing teeth in the maxillary area, seeking for implant therapy.
* Men/Women
* In good systemic health (ASA I/ II)
* Present with no contra indication against oral surgical interventions
* Patients required replacement of a single missing tooth. The tooth at the implant site(s) must have been extracted or lost at least 12 weeks before the date of implantation.
* At least 10 mm of bone in the vertical dimension
* At least 6 mm of bone in the bucco-lingual dimension.
* No need for bone augmentation procedure in any of the dimensions
* Full mouth plaque score (FMPI) lower or equal than 25%

Exclusion Criteria:

* Autoimmune disease require medical treatment
* Medical conditions requiring prolonged use of steroids
* Use of Bisphosphonate intravenously or more then
* Infection (local or systemic) - patient with gingivitis or active local infection will undergo a medical treatment prior to his entrance to the study, each individual will be evaluated prior to study procedure for suitability, in case of systemic infection the evaluation will be based on medical anamneses, and if necessary will be referred to relevant medical tests.
* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Immunocompromised patients
* Uncontrolled Diabetes
* Smokers
* Prisoners

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Fit of the crowns | 1 year
  To measure this parameter we will focus on interproximal fit and occlusion. Interproximal contact points will be checked with dental floss.

SECONDARY OUTCOMES:
Time consumption at the dental chair | 1 year
  Numbers of appointment needed for each procedure will be counted and each one of them will be timed (from the unscrewing of the healing abutment until its replacement).
Time consumption in the lab | 1 year
  The time needed by the lab for manufacturing the crowns will be evaluated by timing all the different steps.
Global cost | 1 year
  Considering the time spent by the dentist and the lab technician, the cost of the optical impression system, of impression materials, of impression trays, of scan bodies and of impression copings, the final cost of each crown will be compared.
Esthetical aspect | 1 year
  A VAS evaluation of the esthetic properties (scoring from zero to ten each crown) will be achieved after the placement of each crown.
Patient centered outcomes | 1 year
  A questionnaire based on VAS scales will be given out and filled by the patients. Thus it will be possible to estimate which of both impressions is less unpleasant for them (questionnaire are in developement).